CLINICAL TRIAL: NCT01276977
Title: Zolmitriptan Nasal Spray VS Eletriptan in the Acute Treatment of Migraine
Brief Title: Zolmitriptan Nasal Spray Versus Eletriptan in the Acute Treatment of Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California Medical Clinic for Headache (Other)
Responsible Party: David Kudrow, M.D., California Medical Clinic for Headache
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRUSZOLM0028
Record Dates: First submitted 2011-01-11; First posted 2011-01-14 (Estimated); Last update posted 2011-01-14 (Estimated); Status verified 2011-01

CONDITIONS: Acute Migraine; Migraine Headache; Headache Disorders
Keywords: Migraine; Acute Migraine; Headache
MeSH Terms: conditions — Migraine Disorders; Headache Disorders; Headache | interventions — zolmitriptan; Nasal Sprays; eletriptan; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zolmitriptan 5 mg nasal spray (Experimental)
  Interventions: Drug: Zolmitriptan 5 mg Nasal Spray; Drug: Eletriptan 40 mg tablet
- Eletriptan 40 mg Tablet (Active Comparator)
  Interventions: Drug: Zolmitriptan 5 mg Nasal Spray; Drug: Eletriptan 40 mg tablet

INTERVENTIONS:
Drug: Zolmitriptan 5 mg Nasal Spray — Patients will treat 2 migraine attacks with zolmitriptan 5 mg nasal spray and 2 migraine attacks with eletriptan.
Drug: Eletriptan 40 mg tablet — Patients will treat 2 migraine attacks with Eletriptan and 2 migraine attacks with zolmitriptan 5 mg nasal spray

SUMMARY:
The purpose of this study is to Compare the efficacy of zolmitriptan 5 mg nasal spray vs. eletriptan 40 mg tablet in the acute treatment of migraine.

To develop and evaluate a set of importance weights for a predefined set of treatment attributes for migraine suffers using zolmitriptan 5 mg nasal spray vs. eletriptan 40 mg tablet.

To contrast the efficacy of zolmitriptan 5 mg nasal spray vs. eletriptan 40 mg tablet at early time points.

To analyze the patterns of self-reported tolerability of migraine sufferers using zolmitriptan 5 mg nasal spray vs. eletriptan 40 mg tablet.

DETAILED DESCRIPTION:
An open-label, randomized, cross-over study comparing the efficacy of zolmitriptan 5 mg nasal spray with eletriptan 40 mg tablet at early time points. Satisfaction endpoints include global assessment of preference, overall satisfaction and effectiveness as well as tolerability of both medications.

ELIGIBILITY:
Inclusion Criteria:

* 15 to 70 years old
* Migraine attacks according to the criteria proposed by the IHS
* 3-12 Migraine attacks per month
* adequate contraception
* Willing and able to give written informed consent
* Willing and able to complete the entire course of the study & comply with instructions
* Stable dose of preventive medication for at least 4 weeks

Exclusion Criteria:

* Disorders listen in groups 5-11 of the IHS Classification
* Subject is pregnant or lactating.
* Significant medical or psychiatric disease
* Subject has a history of symptoms suggestive of ischemic heart disease (angina, myocardial infarction, documented silent ischemia) or other vascular disease, including Prinzmetal angina, claudication, Wolff-Parkinson-White syndrome, or other cardiac accessory conduction pathway arrhythmia
* Subject has uncontrolled hypertension.
* Subject has history of basilar, ophthalmoplegic, or hemiplegic migraine or serious neurologic condition associated with headache
* Subject has used monoamine oxidase A inhibitors (MAOI-As) within 2 weeks of randomization
* Subject has had serious adverse event while using another 5-HT agonist, or previous serious adverse event while using zolmitriptan or hypersensitivity to zolmitriptan or eletriptan
* Using CYP3A4 inhibitors listed by the FDA as contraindicated with eletriptan
* Moderate/severe hepatic/renal impairment
* Subject currently using cimetidine
* Concomitant medication treatment with a triptan, ergotamine or methysergide.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Reduction of migraine headache pain from mild, moderate or severe to pain free. | 30 minutes post-dose

SECONDARY OUTCOMES:
Reduction of migraine headache pain from mild, moderate or severe to pain free. | 15 minutes post-dose

CONTACTS AND LOCATIONS:
Overall Officials: David B Kudrow, MD, Principal Investigator — California Medical Clinic for Headache
Locations (1):
- California Medical Clinic for Headache, Santa Monica, California, United States